CLINICAL TRIAL: NCT01640067
Title: Intra-spinal Cord Delivery of Human Neural Stem Cells in ALS Patients: Proposal for a Phase I Study/ Trapianto Intramidollare di Cellule Staminali Neurali Umane Come Terapia Putativa Per la SLA: Proposta di un Trial Clinico di Fase I
Brief Title: Human Neural Stem Cell Transplantation in Amyotrophic Lateral Sclerosis (ALS)
Acronym: hNSCALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azienda Ospedaliera Santa Maria, Terni, Italy (Other)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other); Università di Padova Italy (Unknown)
Responsible Party: Principal Investigator, Angelo Luigi Vescovi, Scientific Director of Laboratorio Cellule Staminali, Cell Factory e Biobanca AOSP di Terni, Scientific Director IRCCS Casa Sollievo della Sofferenza S.Giovanni Rotondo Italy, Azienda Ospedaliera Santa Maria, Terni, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: EudraCT: 2009-014484-39
Record Dates: First submitted 2012-07-09; First posted 2012-07-13 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; motor neuron disease; stem cells; safety; ALS-FRS-Functional scale R and FVC (%) variation; Survival analysis; Changes in quality of life scales
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human Neural Stem Cells Suspension (Experimental): 50,000 cells/µl. Patients received either unilateral or bilateral hNSCs microinjections (3 microinjections on each side) into the lumbar spinal cord. Each microinjection consisted of 15 µl of the above 50,000cells/µl suspension, yielding a total of 750,000 cells per injection site.
  Interventions: Biological: Human Neural Stem Cells

INTERVENTIONS:
Biological: Human Neural Stem Cells — Surgical microinjection of human neural stem cells on spinal cord of ALS patients
  Other Names: Human Neural Stem Cells Suspension

SUMMARY:
Primary aim of the trial

1. to verify safety and tolerability of expanded human fetal neural stem cells
2. to verify safety and tolerability of a microsurgery human fetal neural stem cells transplantation model
3. to recognize each change in patient's quality of life

Secondary aim of the trial

1. assessment of the impact of human neural stem cells transplantation on the disability of ALS in a clinically significant and measurable way
2. Assessment of the impact of human neural stem cells transplantation on mortality (all causes)

DETAILED DESCRIPTION:
18 patients diagnosed as definite ALS according to the El Escorial criteria will be recruited during two years. The patients will be divided into 3 groups with different severity. Each group will be less compromised than the group that went before them. Their breathing measurements must be at least 60%. Subjects will receive injections of the human foetal neural stem cells into the spinal cord. A variety of tests and examinations will take place every month for the first year and every three months for the next two in order to monitor the course of the disease and the adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or possible ALS according to revised EL Escorial criteria
* Age: 20-75 years
* documented progression of disease during the last 6 months.
* Absence of concomitant diseases
* Adequate assurances of adherence to protocol
* The patient must be able to communicate verbally or with the use of non-verbal communication system

Group 1

* maximum score of 1 on walking item of ALS functional rating scale
* forced vital capacity > or equal to 60

Group 2

* forced vital capacity > or equal to 60
* ambulation difficulties (maximum score of 2 on walking item of ALS functional rating scale)

Group 3

* Independent ambulation (score 4 on a scale ALS-FRS)
* forced vital capacity > or equal to 70

Exclusion Criteria:

The presence of at least one of the following will lead to patient exclusion.

1. psychiatric diseases or other neurological diseases different from ALS
2. other systemic diseases
3. Neoplasms or other diseases reducing life expectancy
4. Antecedent polio infection
5. corticosteroids, immunoglobulin or immunosuppressive treatment
6. involvement in other clinical trials
7. 2 or more critical items in MMPI
8. neuropsychological evaluation suggestive of mental deterioration or cognitive sphere disturbance.
9. Impediments to MRI
10. patients unable to understand informed consent form and study aims.
11. women who are pregnant or childbearing potential for the duration of the study. Non-pregnant status will be documented by beta-HCG negative test 7 days before treatment start

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
safety of a microsurgery human neural stem cells transplantation into spinal cord of ALS patients | Participants will be followed for at least 3 years. Monthly in the first year and every three months the following two years
  * Percentage of subjects (%) with treatment-related mortality defined as death due to procedure and not to the course of the disease
  * Number of adverse events related to the procedure
  * Changes in neuroradiological (MRI) and neurophysiological variables (SEP, MEP)
  * Changes in neuropsychological variables

CONTACTS AND LOCATIONS:
Overall Officials: Angelo L Vescovi, Professor, Principal Investigator — IRCCS Casa Sollievo della Soffernza and AOSP Terni, Italy
Locations (1):
- Azienda Ospedaliera Santa Maria, Terni, Terni, Italy

REFERENCES:
- [Background] Gelati M, Profico D, Projetti-Pensi M, Muzi G, Sgaravizzi G, Vescovi AL. Culturing and expansion of "clinical grade" precursors cells from the fetal human central nervous system. Methods Mol Biol. 2013;1059:65-77. doi: 10.1007/978-1-62703-574-3_6. PMID 23934834
- [Result] Mazzini L, Gelati M, Profico DC, Sgaravizzi G, Projetti Pensi M, Muzi G, Ricciolini C, Rota Nodari L, Carletti S, Giorgi C, Spera C, Domenico F, Bersano E, Petruzzelli F, Cisari C, Maglione A, Sarnelli MF, Stecco A, Querin G, Masiero S, Cantello R, Ferrari D, Zalfa C, Binda E, Visioli A, Trombetta D, Novelli A, Torres B, Bernardini L, Carriero A, Prandi P, Servo S, Cerino A, Cima V, Gaiani A, Nasuelli N, Massara M, Glass J, Soraru G, Boulis NM, Vescovi AL. Human neural stem cell transplantation in ALS: initial results from a phase I trial. J Transl Med. 2015 Jan 27;13:17. doi: 10.1186/s12967-014-0371-2. PMID 25889343
- [Derived] Gelati M, Profico DC, Ferrari D, Vescovi AL. Culturing and Expansion of "Clinical Grade" Neural Stem Cells from the Fetal Human Central Nervous System. Methods Mol Biol. 2022;2389:57-66. doi: 10.1007/978-1-0716-1783-0_5. PMID 34558001
- [Derived] Robberecht W, Philips T. The changing scene of amyotrophic lateral sclerosis. Nat Rev Neurosci. 2013 Apr;14(4):248-64. doi: 10.1038/nrn3430. Epub 2013 Mar 6. PMID 23463272
- See also: No profit Association that grant this study — http://www.revertonlus.org/